CLINICAL TRIAL: NCT00522782
Title: Phase IV Study of the Effect of Nebulized Budesonide on Exhaled Nitric Oxide in Children, Four to Six Years of Age, With Asthma
Brief Title: Effect of Budesonide on Exhaled Nitric Oxide in Asthmatic Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AAADRS Clinical Research Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Miguel Lanz, MD, AAADRS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRUSBUPR-0062
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Active Comparator): Nebulized budesonide
  Interventions: Drug: Nebulized Budesonide; Device: Nitric Oxide Analyzer

INTERVENTIONS:
Drug: Nebulized Budesonide — Pulmicort Respules 0.5mg/2cc
  Other Names: Pulmicort Respules 0.5mg/2ml nebulized
Device: Nitric Oxide Analyzer — Niox NO analyzer
  Other Names: Niox NO analyzer

SUMMARY:
To study the improvement in airway inflammation in children with asthma non-invasively with exhaled breath NO, a marker of inflammation, after therapy with nebulized budesonide as 0.5mg daily.

DETAILED DESCRIPTION:
Comparisons will be made before and after 2 week therapy of nebulized budesonide in children not on prior anti-inflammatory medications.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis previously for 6 months
* Past asthma medication without change for previous 6 months
* Increased NO levels and ability to perform maneuver
* ICF signed by parents

Exclusion Criteria:

* Systemic steroids in past 60 days,inhaled/nebulized steroids in past 4 weeks
* Hospitalization within 3 months
* Upper or lower airways active infection or cigarette smoke direct exposure
* Use of other asthma medications other than bronchodilators one month prior and during the trial
* Noncompliance

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Exhaled breath nitric oxide pre- to post treatment | two weeks

SECONDARY OUTCOMES:
Spirometry with peak flow measurements and daily diary scores | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miguel J Lanz, MD, Principal Investigator — Principal Investigator
Locations (1):
- AAADRS Clinical Research Center, Coral Gables, Florida, United States